CLINICAL TRIAL: NCT03487510
Title: Dysphagia on the Intensive Care Unit - a Multinational European Analysis
Brief Title: Dysphagia on the Intensive Care Unit
Acronym: DICE-SWISS
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Jörg Schefold, Sponsor-investigator, Insel Gruppe AG, University Hospital Bern
Other Study IDs: DICE
Record Dates: First submitted 2018-03-09; First posted 2018-04-04 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2018-05

CONDITIONS: Deglutition Disorders
Keywords: treatment standards; diagnostical approaches; descriptive
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- NO groups: no groups apply.
  Interventions: Other: NO interventions apply

INTERVENTIONS:
Other: NO interventions apply — does not apply

SUMMARY:
Recording of routine practice patterns to detect and/or treat Dysphagia on the ICU via interview of local colleagues. This will not allow to record generalizable data, but will reflect the actual routine standard of care.

ELIGIBILITY:
Inclusion criteria:

* All senior ICU physicians in charge for adult critically ill ICU patients. Respective ICUs must be accredited by the "Schweizerische Gesellschaft für Intensivmedizin".
* ICUs located in Switzerland.
* Senior ICU physicians willing to voluntarily fill in the provided questionnaire.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Senior local ICU physicians (Swiss ICUs only).
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2017-11-11 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Number of centers using fibre-optic endoscopic evaluation of swallowing (FEES) vs. non-instrumental methods to detect/ treat dysphagia on the ICU. | through study completion, an average of 1 month
  Analysis of number of ICUs using instrumental methods (FEES) vs. non-instrumental methods in local (Swiss) centers to detect dysphagia in the ICU.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Zürcher, MD, Principal Investigator — Inselspital, University of Bern
Locations (1):
- Dept. of Intensive Care Medicine, University of Bern,, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No